CLINICAL TRIAL: NCT04955054
Title: the Association of Intestinal Microbial Metabolites and Cardiac Function in Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020362
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Acute Myocardial Infarction
Keywords: bile acids; short chain fatty acid; cardiac function
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: patients without coronary artery disease
- UAP: patients without unstable angina pectoris
  Interventions: Diagnostic Test: diagnose
- AMI: patients with acute myocardial infarction
  Interventions: Diagnostic Test: diagnose

INTERVENTIONS:
Diagnostic Test: diagnose — Patients from UAP and AMI meet the criteria of UAP or STEMI.
  Groups: AMI; UAP

SUMMARY:
Recently, more and more studies have confirmed that intestinal flora is closely related to the occurrence and development of cardiovascular diseases.Bile acids (BAS), short chain fatty acids (SCFA) and trimethylamine oxide (TMAO), the main metabolites of intestinal flora, are the key mediators of the interaction between gut and host. We aim to explore the association of BAs and SCFA with cardiac function in patients with AMI.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in China, and acute myocardial infarction (AMI) is the main cause of death of cardiovascular disease. In recent years, clinical epidemiological studies have confirmed that intestinal flora is closely related to the occurrence and development of cardiovascular diseases such as diabetes, hyperlipidemia, hypertension, atherosclerosis, coronary heart disease, heart failure and so on. Bile acids (BAS), short chain fatty acids (SCFA) and trimethylamine oxide (TMAO), the main metabolites of intestinal flora, are the key mediators of the interaction between gut and host. It is suggested that intestinal flora and its metabolites participate in the pathophysiological process of cardiovascular disease through inflammation, oxidative stress and programmed death, and have the potential to be intervention targets. Basic and clinical studies have shown that TMAO is associated with the onset and poor prognosis of AMI by promoting the development of atherosclerosis and thrombosis, but there are few reports on the relationship between BAs or SCFA and AMI. We aim to explore the association of BAs and SCFA with cardiac function in patients with AMI.

ELIGIBILITY:
Inclusion Criteria:

The patient, aged 18-85 years, had undergone coronary angiography and agreed to be enrolled and signed the informed consent.

AMI : according to ST segment elevation myocardial infarction diagnostic criteria.

UAP:

1. typical chest pain symptoms;
2. negative in markers of myocardial injury;
3. The stenosis of main coronary artery or its main branches is more than 50%

Control:

1. atypical chest pain symptoms
2. negative in markers of myocardial injury;
3. The stenosis of main coronary artery and its main branches is less than 50%

Exclusion Criteria:

1. Acute infection or application of antibiotics in the past 3 months;
2. Chronic heart failure;
3. History of inflammatory or absorptive bowel disease and bowel resection;
4. Acute, chronic liver disease or other reasons lead to abnormal liver function (transaminase is more than 5 times of normal value);
5. Renal insufficiency (serum creatinine > 220μml/L or creatinine clearance rate < 30 ml/min);
6. Malignant tumor;
7. Autoimmune diseases;
8. Uninformed patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient, aged 18-85 years, had undergone coronary angiography and agreed to be enrolled and signed the informed consent. And they met the inclusion criteria and did not meet the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-11 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the plasma levels of BAs and SCFA | one week
  the plasma levels of bile acids and short chain fatty acid in fast

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No